CLINICAL TRIAL: NCT03027219
Title: Prospective Observational Study of the Changes of Blood Flow of Arterial Anastomosis-site of Free Flap in Diabetic Patients Who Undergoing Free Flap Transfer
Brief Title: Blood Flow Change After Free Flap Surgery in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, Professor, Asan Medical Center
Other Study IDs: S2016-2043-0003
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Alprostadil

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Alprostadil — Vasodilator for anastomosis-site of free flap
  Other Names: Eglandin

SUMMARY:
We aim to evaluate the flow change of arterial anastomosis site during free flap surgery in diabetic patients.

DETAILED DESCRIPTION:
Objective: flow change of arterial anastomosis site during free flap surgery in diabetic patients.

Background: No research was published about flow change of arterial anastomosis site of the free flap during surgery.

Plan: Using Duplex sonography, various parameters related flap perfusion will be evaluated before and after the administration of alprostadil.

ELIGIBILITY:
Inclusion Criteria:

1. Plan to receive free flap transfer under general anesthesia
2. Age: >=18 and <80 years old
3. History of diabetes mellitus
4. Administration of alprostadil during surgery
5. Volunteer, who are provided written informed consent prior to study participation

Exclusion Criteria:

1. Refuse the participation of study
2. >= American society of anesthesiologist physical status IV
3. Use of any vasopressor or inotropic for hemodynamic instability before participation of study
4. Inappropriate subjects who are identified by researchers

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients who are undergoing free flap surgery
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
Flow change | before alprostadil administration, 30 mins after alprostadil administration
  Peak velocity of anastomosis-site of free flap

CONTACTS AND LOCATIONS:
Overall Officials: Young-kug Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No